CLINICAL TRIAL: NCT05268276
Title: The Effect of Designed Protocol of Care on the Outcomes of Postpartum Perineal Trauma: a Randomized Controlled Trial (RCT)
Brief Title: Designed Protocol of Care for Postpartum Perineal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asmaa Abdallah Ahmed Hussein (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Asmaa Abdallah Ahmed Hussein, assisstant lecturer at faculty of nursing /cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asmaa Abdallah Ahmed Hussein
Record Dates: First submitted 2021-12-27; First posted 2022-03-07 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Perineal Injury
Keywords: perineal trauma; outcomes; pospartum; protocol of care

STUDY DESIGN:
Intervention Model Description: after obtaining the primary and official permission data collection will be carried out through five steps in each group: Recruitment & randomization; interviewing; initial assessment; intervention; follow up and monitoring. : For the study group the intervention will be according to a designed protocol of care that entails; 1) Application of ice gel pad on perineal trauma for the first 24 hours post partum; 2) Performance of pelvic floor exercises (Kegel exercises) from six hours till one week postpartum; 3) Application of warm compresses after 48 hours and through the first week postpartum. The investigator will perform demonstration and then redemonstration by the women on each intervention will be done. A designed booklet (developed previously) that explains each intervention will be given to each woman.The control group will receive the routine hospital care only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group will recelve adesigned protocol of care that entails three interventions as the following1) Application of ice gel pad on perineal trauma for the first 24 hours post partum 2) Performance of pelvic floor exercises (Kegel exercises) from six hours till one week postpartum 3) Application of warm compresses after 48 hours and through the first week postpartum.
  The investigator will perform demonstration and then redemonstration by the women on each intervention will be done. A designed booklet (developed previously) that explains each intervention will be given to each woman.
  Interventions: Other: 1-perineal ice-gel pad application; Other: 2-performance of pelvic floor exercises (Kegel exercises); Other: 3- perineal warm compresses application
- control group (No Intervention): The control group will receive the routine hospital care only

INTERVENTIONS:
Other: 1-perineal ice-gel pad application — For the study group Immediately after delivery (within 30 minutes to one hour after delivery), an ice gel pad will be applied to perineal trauma. each gel pad will have fixed standardized diameter (an approximately 5 cm width, 23 cm length, and 1.5 cm thickness) and approved by Egyptian ministry of health. It will be kept in the freezer for 45-60 minutes and will be removed when frozen. Then, it will be wrapped in a sterile pad and applied to cover the perineum and anal region.The investigator will provide a clear and concise information through oral and written instructions about the following; 1) The ice gel pad's purpose, benefits, anticipated effects and how to apply it, 2) Apply the ice gel pad on perineum after birth within 30 minutes to an hour, 3) Instruct the women to apply the ice gel pad for about 20 minutes every two hours during the first 24 hours postpartum only
  Arms: study group
Other: 2-performance of pelvic floor exercises (Kegel exercises) — women will receive instructions to practice pelvic floor exercises (Kegel exercises) and will be asked to perform these exercises from 6 hours postpartum and continue at home till one week. Before applying the technique, the investigator will teach the women how to recognize the accurate muscle, whereby she imagines holding passing gases or trying to stop the flow of urine midstream at the same time. The women will be taught to insert a clean finger into the vagina before practicing the exercises and if the women feeling pressure around her finger, she is on the right track, . The investigator will perform vaginal examination while the woman is doing the pelvic floor exercises (Kegel exercises) to ensure correct use of muscles. The investigator will instruct the women to continue contracting the muscles for about 5 seconds and then to loosen them for 5 seconds and repeat it for five times each set, perform at least five sets per day
  Arms: study group
Other: 3- perineal warm compresses application — women will be instructed to apply warm compresses on perineal trauma 48 hours postpartum at home. This will be done by using a clean pad soaked in warm water and squeezed to remove excess water then placed gently on the perineum, the warm compresses will be applied for 15 minutes three times per day (every 8 hours), and water in the bowl will be replaced with every application. Women will be asked to apply warm compresses on perineal trauma from 48 hours postpartum till one week.
  Arms: study group

SUMMARY:
the study is intended to test the effect of designed protocol of care that include perineal ice-gel pad application, performance of pelvic floor exercises (Kegel exercises) and perineal warm compresses application on the outcomes of postpartum perineal trauma among women with vaginal delivery at postpartum ward.To fulfill the aim of this study the following research hypothesis is formulated: H1: Post partum women with perineal trauma who will receive the designed protocol of care will have better perineal trauma outcomes than those who will receive the routine hospital care.Sub-hypothesis 1: Postpartum women with perineal trauma who will receive the designed protocol of care will show better perineal trauma healing than those who will receive the routine hospital care.

Sub-hypothesis 2: Postpartum women with perineal trauma who will receive the designed protocol of care will have less perineal pain score than those who will receive the routine hospital care.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted to test the effect of designed protocol of care that include; perineal ice-gel pad application for the first 24 hours after delivery, performance of pelvic floor exercises (Kegel exercises) for six hours till one week postpartum and perineal warm compresses application from 48 hours till one week postpartum on the outcomes of postpartum perineal trauma .The study will be conducted on (100) postpartum women with normal spontaneous vaginal delivery and having postpartum perineal trauma that randomly assigned to either study group (50) women or control group (50) women.The study will be conducted at postpartum ward of emergency department for labor and delivery in Obstetrics and Gynecology Hospital at Kasr El Aini University Hospital affiliated to Cairo University.Required data will be collected by using 5 tools: A) Structured interview schedule; B) Visual Analogue Scale for pain intensity(VAS); C) Visual Analogue Scale (VAS) for rating functional activities; D) Standardized REEDA scale; and E) Postpartum follow up sheet. the primary official permission will be obtained from the research ethics committee of faculty of nursing, Cairo University to approve the tools and the study. An official permission will be granted from the hospital administrative personnel in the recommended setting to collect the data. Then, data collection will be carried out through five steps in each group: Recruitment & randomization; interviewing; initial assessment; intervention; follow up and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be according to the following

  1. primiparous or 2nd. multiparaous women with postpartum perineal trauma either episiotomy or perineal tear (first and second degree only)
  2. age not exceeding 40 years
  3. body mass index (BMI)within normal 18.5-24.9 kg/m2 or overweight 25-29.9 kg/m2,
  4. free from any high risk condition affecting perineal trauma healing (e.g., diabetes mellitus or obesity),
  5. over 37 week gestation
  6. not having any complications during labor and delivery(e.g., abnormal presentation, obstructed labor or delivered with instrument),
  7. not having any immediate postnatal complications such as postpartum hemorrhage.

Exclusion Criteria:

1. 3rd or 4th degree perineal tear
2. obesity.
3. age more than 40 years
4. having any complications during labor and delivery(e.g., abnormal presentation, obstructed labor or delivered with instrument)
5. having any immediate postnatal complications such as postpartum hemorrhage. ]

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdallah, Principal Investigator — Cairo University; Yousria Ahmed, Study Director — Cairo University; Shadia Abdel Kader, Study Director — Cairo University
Locations (1):
- faculty of nursing/Cairo university& Kasr El Aini University Hospital, Cairo, El-manial, Egypt

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: no participants were excluded for the study after enrollment and before assignment to study or control group
Groups:
- Study Group: Intervention for the study group was carried out according to a designed protocol of care that entails: 1) application of an ice gel pad on perineal trauma for 20 minutes every two hours during the first 24 hours postpartum; 2) performance of pelvic floor exercises (Kegel exercises) five times daily starting from six hours till one week postpartum; and 3) application of warm compresses for 15 minutes three times daily starting after 48 hours and through the first week postpartum. On each intervention, the investigator demonstrated and then redemonstrated with the women. A specially designed booklet (developed previously) that explains each intervention was given to each woman.
- Control Group: the control group received the routine hospital care (antibiotic every 12 hours and analgesic as needed )
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 50 | 50
Completed | 47 | 45
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control Group: The control group received the routine hospital care only
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants] — the age of participants included at the study was from 18-40 years
  Participants
    Age: 18-20 years | 12 | 9 | 21
    Age: 21-30 years | 28 | 32 | 60
    Age: 31-40 years | 10 | 9 | 19
Sex/Gender, Customized [Count of Participants; unit: Participants]
  gender: female | 50 | 50 | 100
  gender: male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
level of education [Count of Participants; unit: Participants]
  Read &Write | 10 | 8 | 18
  Primary School | 3 | 11 | 14
  Preparatory School | 14 | 8 | 22
  Secondary School | 16 | 17 | 33
  University School | 7 | 6 | 13
occupation [Count of Participants; unit: Participants]
  House wife | 46 | 45 | 91
  Working | 4 | 5 | 9
residence [Count of Participants; unit: Participants]
  Rural | 14 | 16 | 30
  Urban | 36 | 34 | 70
gravidity [Count of Participants; unit: Participants] — primigravida : women who is pregnant on time gravida 2: women who is pregnant 2 times gravida 3: women who is pregnant 3 times gravida 4: women who is pregnant 4 times
  Participants
    Primi gravida | 22 | 13 | 35
    Gravida 2 | 17 | 23 | 40
    Gravida 3 | 9 | 9 | 18
    Gravida 4 | 2 | 5 | 7
Body Mass Index(BMI) [Count of Participants; unit: Participants] — normal weight: when BMI between (18.5- 24.9 kg/m2 ), overweight : when BMI between (25- 29.9 kg/m2)
  Participants
    Normal | 30 | 33 | 63
    Over weight | 20 | 17 | 37
type of perineal trauma [Count of Participants; unit: Participants]
  Episiotomy | 45 | 42 | 87
  Perineal tear | 2 | 4 | 6
  both episiotomy and perineal tear | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Severity of Postpartum Perineal Pain
Description: Postpartum severity of perineal pain will be assessed by Visual Analogue Scale for pain intensity (VAS).It is a self-reported 10 cm horizontal line which represents the subjective estimation of pain intensity. It comprises 0-10-point numerical scale, the two opposite ends representing no pain to severe pain as follows: no pain (0), mild pain (< 4), moderate pain (4 - < 8), and sever pain (8-10).
Time Frame: one hour after delivery, six hours after delivery, 24 hours after delivery, day 3 after delivery, day 5 after delivery, day 7 after delivery
Population: severity of postpartum perineal pain
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: The control group received the routine hospital care
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  one hour after delivery | 8.200 (1.21) | 8.280 (1.27)
  six hours after delivery | 4.500 (1.87) | 8.080 (1.17)
  24 hours after delivery | 3.880 (2.12) | 8.020 (.97)
  day 3 after delivery | 2.520 (1.94) | 7.720 (1.16)
  day 5 after delivery | 1.260 (2.26) | 4.700 (2.05)
  day 7 after delivery | .7800 (2.15) | 2.46 (2.64)

2. Primary Outcome: Postpartum Perineal Trauma Healing
Description: Postpartum perineal trauma healing will be assessed by standardized Redness,Edema,Echymosis,Discharge,Approximation of sutures( REEDA) scale.The total score ranged from 0 to 15 and categorized as the following; 0 to 2 good wound healing , 3 to 5 moderate wound healing, 6 to 8 mild wound healing, and 9 to 15 poor wound healing . the lower score 0 and the maximum score 15 , as the score decreases it indicate better wound healing
Time Frame: one hour after delivery, six hours after delivery, day 7after delivery
Population: severity of postpartum perineal pain
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  one hour after delivery | 9.240 (1.91) | 9.14 (1.94)
  6 hours after delivery | 6.460 (2.09) | 9.04 (1.88)
  day 7 after delivery | .740 (1.41) | 1.78 (1.56)

3. Secondary Outcome: Occurrence of Postpartum Perineal Trauma Infection
Description: Postpartum perineal trauma infection will be assessed by standardized REEDA scale.
  the score ranged from 0-15 , score from 0 to 2 indicates no wound infection,while from 3-15 indicates wound infection
Time Frame: day 7 after delivery
Population: postpartum perineal wound infection
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 50 | 50
Participants
  infection | 7 | 13
  no infection | 43 | 37

4. Secondary Outcome: Postpartum Difficulty With Performing Functional Activity
Description: postpartum difficulty with performing functional activity as (turning/rolling in bed, getting out of bed, sitting, walking, defecation and urination) will be assessed using Visual Analogue Scale for rating functional activity.The scoring for each activity will be as follows: no difficulty (0), mild difficulty (< 4), moderate difficulty (4 - <8), and sever difficulty (8-10). The total score will be recorded (0-60 point), the lowest score (0) indicate no difficulties and the maximum score (60) indicate maximum difficulty. The total score will be interpreted as the following no difficulties (0), Mild difficulties (1 - < 24), Moderate difficulties (24 - < 48), Sever difficulties (48-60).
Time Frame: 24 hours after delivery, day 3 after delivery, day 5 after delivery
Population: postpartum difficulties with daily infection
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 50 | 50
Participants
  24 hours after delivery: no difficulty | 0 | 0
  24 hours after delivery: mild difficulty | 5 | 0
  24 hours after delivery: moderate difficulty | 37 | 17
  24 hours after delivery: sever difficulty | 8 | 33
  day 3 after delivery: no difficulty | 9 | 0
  day 3 after delivery: mild difficulty | 34 | 0
  day 3 after delivery: moderate difficulty | 6 | 16
  day 3 after delivery: sever difficulty | 1 | 34
  day 5 after delivery: no difficulty | 31 | 7
  day 5 after delivery: mild difficulty | 15 | 23
  day 5 after delivery: moderate difficulty | 2 | 15
  day 5 after delivery: sever difficulty | 2 | 5

ADVERSE EVENTS:
Time Frame: over one week pospartum
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT05268276/Prot_SAP_000.pdf